CLINICAL TRIAL: NCT01607255
Title: Comparative Efficacy of Water & Indigo Carmine vs Water or Air Method
Brief Title: Comparative Efficacy of Water & Indigo Carmine vs. Water or Air Method on Adenoma Detection Rate (ADR) - a Randomized Controlled Trial (RCT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN-10-11S
Record Dates: First submitted 2012-05-24; First posted 2012-05-30 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Neoplasms
Keywords: adenoma detection; screening colonoscopy; water exchange method; chromoendoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Indigo Carmine; Water; Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- water (exchange) method (Experimental): Residual pocket of air will be suctioned. Water is infused using a peristaltic pump to facilitate scope advancement until the cecum is reached. Dirty water will be suctioned and clean water is infused. Air will not be insufflated until the cecum is reached. Residual water is suctioned and air insufflated on scope withdrawal to facilitate biopsy and removal of lesions.
  Interventions: Procedure: water (exchange) method
- water (exchange) plus dye method (Experimental): Residual pocket of air will be suctioned. Water with 0.008% indigocarmine is infused using a peristaltic pump to facilitate scope advancement until the cecum is reached. Dirty water will be suctioned and clean water is infused. Air will not be insufflated until the cecum is reached. Residual water is suctioned and air insufflated on scope withdrawal to facilitate biopsy and removal of lesions
  Interventions: Drug: Indigo carmine; Procedure: water (exchange) plus dye method
- air method (Active Comparator): The colonoscope is inserted gently and advanced slowly using minimal air insufflation, if necessary, the assistant will provide abdominal compression or the patient's position will be changed to facilitate scope passage. The scope is inserted until the cecum is reached. Air is insufflated on scope withdrawal for visualization and water irrigation is used to remove any adherent feces covering the mucosa. Biopsy or polypectomy is performed where indicated.
  Interventions: Procedure: air method

INTERVENTIONS:
Drug: Indigo carmine — 0.008% indigo carmine in water is used as a surface contrast agent to enhance visualization of diminutive polyps (adenoma) during screening colonoscopy
  Arms: water (exchange) plus dye method
Procedure: water (exchange) method — Residual pocket of air will be suctioned. Water is infused using a peristaltic pump to facilitate scope advancement until the cecum is reached. Dirty water will be suctioned and clean water is infused. Air will not be insufflated until the cecum is reached. Residual water is suctioned and air insufflated on scope withdrawal to facilitate biopsy and removal of lesions.
  Arms: water (exchange) method
Procedure: water (exchange) plus dye method — Residual pocket of air will be suctioned. Water with 0.008% indigocarmine is infused using a peristaltic pump to facilitate scope advancement until the cecum is reached. Dirty water will be suctioned and clean water is infused. Air will not be insufflated until the cecum is reached. Residual water is suctioned and air insufflated on scope withdrawal to facilitate biopsy and removal of lesions
  Arms: water (exchange) plus dye method
Procedure: air method — The colonoscope is inserted gently and advanced slowly using minimal air insufflation, if necessary, the assistant will provide abdominal compression or the patient's position will be changed to facilitate scope passage. The scope is inserted until the cecum is reached. Air is insufflated on scope withdrawal for visualization and water irrigation is used to remove any adherent feces covering the mucosa. Biopsy or polypectomy is performed where indicated.
  Arms: air method

SUMMARY:
Adenoma detection rate (ADR) is a quality indicator of colonoscopy performed for colorectal cancer screening. Population studies have shown that traditional air colonoscopy fails to eliminate post screening colonoscopy cancers or cancer mortality in the proximal colon. The investigators aim to establish the superior effectiveness of combining chromoendoscopy with the water exchange method in detecting more proximal diminutive adenomas during screening colonoscopy in sedated Veterans. An improved adenoma detection rate associated with optical colonoscopy will minimize the risk of missed lesions. The improvement may translate into a remedy for the limitations of screening colonoscopy in the proximal colon, e.g. a higher adenoma detection rate may minimize the burden of post screening colonoscopy interval colorectal cancers among the veteran population.

DETAILED DESCRIPTION:
1. Design: Prospective, single center, patient blinded, randomized controlled trial
2. Methods: Colonoscopy with traditional air insufflation, water exchange or water exchange plus indigocarmine to aid insertion of colonoscope; split dose bowel preparation; all patients will receive sedation; assessment of serum electrolytes level before and after colonoscopy

   1. Control method: Traditional air insufflation method.
   2. Study methods:

      * Water exchange method.
      * Water method combined with chromoendoscopy (0.008% indigo carmine).
3. Population to be studied Veterans between age 50 and 75 referred for first time screening colonoscopy
4. Unit(s) of analysis

   1. Primary outcome: overall adenoma detection rate.
   2. Secondary outcomes: patient demographic variable and procedure related measures.
5. Sampling strategy: all Veterans referred for screening colonoscopy will be offered enrollment in the study.

   1. Sample size calculation. A total of 480 subjects will be recruited and randomized with 160 in each group.

5. Subject recruitment: patients referred for screening colonoscopy come from three sources.

6. Description of base population and groups to be studied and method of randomization.

Veterans between age 50 and 75 referred for first time screening colonoscopy. After informed consent, assignment to control or study arm based on computer generated random number codes stored in pre-arranged opaque envelopes.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic Veterans scheduled for first time screening colonoscopy and agree to be randomized will be enrolled.

Exclusion Criteria:

* patients who decline to be randomized, non screening cases.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2013-05-16 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W. Leung, MD, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leung JW, Ransibrahmanakul K, Toomsen L, Mann SK, Siao-Salera R, Leung FW. The water method combined with chromoendoscopy enhances adenoma detection. J Interv Gastroenterol. 2011 Apr;1(2):53-58. doi: 10.4161/jig.1.2.16827. PMID 21776426
- [Background] Leung FW, Leung JW, Siao-Salera RM, Mann SK, Jackson G. The water method significantly enhances detection of diminutive lesions (adenoma and hyperplastic polyp combined) in the proximal colon in screening colonoscopy - data derived from two RCT in US veterans. J Interv Gastroenterol. 2011 Apr;1(2):48-52. doi: 10.4161/jig.1.2.16826. PMID 21776425
- [Background] Leung JW, Do LD, Siao-Salera RM, Ngo C, Parikh DA, Mann SK, Leung FW. Retrospective analysis showing the water method increased adenoma detection rate - a hypothesis generating observation. J Interv Gastroenterol. 2011 Jan;1(1):3-7. doi: 10.4161/jig.1.1.14585. PMID 21686105
- [Background] Leung J, Mann S, Siao-Salera R, Ransibrahmanakul K, Lim B, Canete W, Samson L, Gutierrez R, Leung FW. A randomized, controlled trial to confirm the beneficial effects of the water method on U.S. veterans undergoing colonoscopy with the option of on-demand sedation. Gastrointest Endosc. 2011 Jan;73(1):103-10. doi: 10.1016/j.gie.2010.09.020. PMID 21184876
- [Background] Leung JW, Mann SK, Siao-Salera R, Ransibrahmanakul K, Lim B, Cabrera H, Canete W, Barredo P, Gutierrez R, Leung FW. A randomized, controlled comparison of warm water infusion in lieu of air insufflation versus air insufflation for aiding colonoscopy insertion in sedated patients undergoing colorectal cancer screening and surveillance. Gastrointest Endosc. 2009 Sep;70(3):505-10. doi: 10.1016/j.gie.2008.12.253. Epub 2009 Jun 24. PMID 19555938
- [Background] Leung JW, Thai A, Yen A, Ward G, Abramyan O, Lee J, Smith B, Leung F. Magnetic endoscope imaging (ScopeGuide) elucidates the mechanism of action of the pain-alleviating impact of water exchange colonoscopy - attenuation of loop formation. J Interv Gastroenterol. 2012 Jul;2(3):142-146. doi: 10.4161/jig.23738. Epub 2012 Jul 1. PMID 23805397
- [Background] Yen AW, Leung JW, Leung FW. A new method for screening and surveillance colonoscopy: Combined water-exchange and cap-assisted colonoscopy. J Interv Gastroenterol. 2012 Jul;2(3):114-119. doi: 10.4161/jig.23730. Epub 2012 Jul 1. PMID 23805389
- [Background] Yen AW, Leung JW, Leung FW. A novel method with significant impact on adenoma detection: combined water-exchange and cap-assisted colonoscopy. Gastrointest Endosc. 2013 Jun;77(6):944-8. doi: 10.1016/j.gie.2013.01.011. Epub 2013 Mar 6. PMID 23473001
- [Background] Leung JW, Siao-Salera R, Abramyan O, Mann SK, Ward G, Yen A, Gutierrez R, Leung FW. Impact of water exchange colonoscopy on serum sodium and potassium levels: an observational study. Dig Dis Sci. 2014 Mar;59(3):653-7. doi: 10.1007/s10620-013-2934-0. Epub 2013 Nov 20. PMID 24254340
- [Background] Ngo C, Leung JW, Mann SK, Terrado C, Bowlus C, Ingram D, Leung FW. Interim report of a randomized cross-over study comparing clinical performance of novice trainee endoscopists using conventional air insufflation versus warm water infusion colonoscopy. J Interv Gastroenterol. 2012 Jul;2(3):135-139. doi: 10.4161/jig.23736. Epub 2012 Jul 1. PMID 23805395
- [Background] Leung J, Mann S, Siao-Salera R, Ngo C, McCreery R, Canete W, Leung F. Indigocarmine added to the water exchange method enhances adenoma detection - a RCT. J Interv Gastroenterol. 2012 Jul;2(3):106-111. doi: 10.4161/jig.23728. Epub 2012 Jul 1. PMID 23805387
- [Background] Leung FW, Pan Y, Mann SK, Leung JW, Siao-Salera RM, Jackson G. The water exchange method and difficult colonoscopy. J Interv Gastroenterol. 2012 Jul;2(3):103-105. doi: 10.4161/jig.23727. Epub 2012 Jul 1. No abstract available. PMID 23805386
- [Result] Leung F, Harker J, Leung J, Siao-Salera R, Mann S, Ramirez F, Friedland S, Amato A, Radaelli F, Paggi S, Terruzzi V, Hsieh Y. Removal of infused water predominantly during insertion (water exchange) is consistently associated with a greater reduction of pain score - review of randomized controlled trials (RCTs) of water method colonoscopy. J Interv Gastroenterol. 2011 Jul;1(3):114-120. doi: 10.4161/jig.1.3.18510. Epub 2011 Jul 1. PMID 22163081

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Water (Exchange) Method | Water (Exchange) Plus Dye Method | Air Method
Started | 161 | 160 | 159
Completed | 161 | 160 | 159
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Water (Exchange) Method | Water (Exchange) Plus Dye Method | Air Method | Total
Number analyzed (Participants) | 161 | 160 | 159 | 480
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 102 | 105 | 106 | 313
  >=65 years | 59 | 55 | 53 | 167
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 24 | 65
  Male | 139 | 141 | 135 | 415
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — The study patients were asked which ethnicity they identified with during the pre-procedure assessment.
  Participants
    Hispanic or Latino | 14 | 12 | 11 | 37
    Not Hispanic or Latino | 146 | 147 | 148 | 441
    Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 161 | 160 | 159 | 480
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (4.1) | 29.2 (4.3) | 29.4 (4.3) | 29.4 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Detected Proximal Diminutive (<10 mm) Adenoma Detection Rate
Description: Proximal diminutive adenoma detection rate (ADR) in screening colonoscopy performed with the unusual air method, versus the water (exchange) method and with dye added to the water (exchange) method
Time Frame: 36 months
Measure: Number; unit: participants
Arm/Group | Water (Exchange) Method | Water (Exchange) Plus Dye Method | Air Method
Number analyzed (Participants) | 161 | 160 | 159
participants
  Proximal ADR | 86 | 89 | 83
  Serrated Lesion | 38 | 42 | 18

ADVERSE EVENTS:
Time Frame: Immediate adverse event data were collected within 7 days and long-term complication data were collected at 30 days.
Arm/Group | Water (Exchange) Method | Water (Exchange) Plus Dye Method | Air Method
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/160 | 0/159
Serious Adverse Events (participants affected / at risk) | 4/161 | 3/160 | 1/159
Other Adverse Events (participants affected / at risk) | 0/161 | 0/160 | 0/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Water (Exchange) Method (N=161) | Water (Exchange) Plus Dye Method (N=160) | Air Method (N=159)
post polypectomy abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
post procedural bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
cardiovascular event (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The limitations and caveat of this clinical study are: single center, single blinded (patients) study, single operator, and Veteran patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT01607255/Prot_SAP_000.pdf